CLINICAL TRIAL: NCT06877208
Title: The Effect of Glucagon on Cerebral Glucose Metabolism in Healthy Humans
Acronym: GluCoMet_CD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolai Jacob Wewer Albrechtsen (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Sponsor-Investigator, Nicolai Jacob Wewer Albrechtsen, Principal Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GluCoMet_pilotCD
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Glucose Metabolism
Keywords: Glucagon; 18F-FDG PET; Quantitative PET; Cerebral Glucose Metabolism; Blood-brain Glucose Transfer
MeSH Terms: interventions — Glucagon; Glucose Clamp Technique; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Acute effect (part C): Glucagon, Saline and Glucose Clamp (Experimental): The arm includes three study days. Study day sequence: Glucagon, Saline and Glucose clamp.
  An 18F-FDG PET scan will be performed approximately 15-55 minutes after infusion start.
  Interventions: Other: Glucagon (part C); Other: Glucose clamp (part C); Other: Saline (part C)
- Acute effect (part C): Saline, Glucagon and Glucose Clamp (Experimental): The arm includes three study days. Study day sequence: Saline, Glucagon and Glucose clamp.
  An 18F-FDG PET scan will be performed approximately 15-55 minutes after infusion start.
  Interventions: Other: Glucagon (part C); Other: Glucose clamp (part C); Other: Saline (part C)
- Acute effect (part C): Glucagon, Glucose Clamp and Saline (Experimental): The arm includes three study days. Study day sequence: Glucagon, Glucose clamp and Saline.
  An 18F-FDG PET scan will be performed approximately 15-55 minutes after infusion start.
  Interventions: Other: Glucagon (part C); Other: Glucose clamp (part C); Other: Saline (part C)
- Later effect (part D): Glucagon, Saline and Glucose Clamp (Experimental): The arm includes three study days. Study day sequence: Glucagon, Saline and Glucose clamp.
  An 18F-FDG PET scan will be performed approximately 150-190 minutes after infusion start.
  Interventions: Other: Glucagon (part D); Other: Glucose clamp (part D); Other: Saline (part D)
- Later effect (part D): Saline, Glucagon and Glucose Clamp (Experimental): The arm includes three study days. Study day sequence: Saline, Glucagon and Glucose clamp.
  An 18F-FDG PET scan will be performed approximately 150-190 minutes after infusion start.
  Interventions: Other: Glucagon (part D); Other: Glucose clamp (part D); Other: Saline (part D)
- Later effect (part D): Glucagon, Glucose Clamp and Saline (Experimental): The arm includes three study days. Study day sequence: Glucagon, Glucose clamp and Saline.
  An 18F-FDG PET scan will be performed approximately 150-190 minutes after infusion start.
  Interventions: Other: Glucagon (part D); Other: Glucose clamp (part D); Other: Saline (part D)

INTERVENTIONS:
Other: Glucagon (part C) — 90 minutes intravenous infusion with glucagon (infusion rate of 10 ng/kg/min).
  Arms: Acute effect (part C): Glucagon, Glucose Clamp and Saline; Acute effect (part C): Glucagon, Saline and Glucose Clamp; Acute effect (part C): Saline, Glucagon and Glucose Clamp
Other: Glucose clamp (part C) — 90 minutes intravenous infusion of 20 % weight/volume glucose (in an ajustable rate to match the glucose levels achieved during the glucagon infusion).
  Arms: Acute effect (part C): Glucagon, Glucose Clamp and Saline; Acute effect (part C): Glucagon, Saline and Glucose Clamp; Acute effect (part C): Saline, Glucagon and Glucose Clamp
Other: Saline (part C) — 90 minutes intravenous infusion with isotonic NaCl.
  Arms: Acute effect (part C): Glucagon, Glucose Clamp and Saline; Acute effect (part C): Glucagon, Saline and Glucose Clamp; Acute effect (part C): Saline, Glucagon and Glucose Clamp
Other: Glucagon (part D) — 210 minutes intravenous infusion with glucagon (infusion rate of 10 ng/kg/min).
  Arms: Later effect (part D): Glucagon, Glucose Clamp and Saline; Later effect (part D): Glucagon, Saline and Glucose Clamp; Later effect (part D): Saline, Glucagon and Glucose Clamp
Other: Glucose clamp (part D) — 210 minutes intravenous infusion of 20 % weight/volume glucose (in an ajustable rate to match the glucose levels achieved during the glucagon infusion).
  Arms: Later effect (part D): Glucagon, Glucose Clamp and Saline; Later effect (part D): Glucagon, Saline and Glucose Clamp; Later effect (part D): Saline, Glucagon and Glucose Clamp
Other: Saline (part D) — 210 minutes intravenous infusion with isotonic NaCl.
  Arms: Later effect (part D): Glucagon, Glucose Clamp and Saline; Later effect (part D): Glucagon, Saline and Glucose Clamp; Later effect (part D): Saline, Glucagon and Glucose Clamp

SUMMARY:
This is a pilot study in which the investigators will investigate the effect of exogenous glucagon on cerebral glucose metabolism in healthy humans.

Participants will participate in either part C or part D of the study, and each participant will participate in three study days. During a study day the participant will receive an intravenous infusion of either glucagon, glucose (in an adjustable rate to match to glucose concentrations achieved with the glucagon infusion) or saline. During each study day an 18F-flouro-deoxy-glucose (FDG) Positron Emission Tomography (PET)/Computed Tomography (CT) scan will be performed to quantify cerebral glucose metabolism during the first part (acute effect) of the glucagon/glucose/saline infusion (part C) or the last part (later effect) of the glucagon/glucose/saline infusion (part D).

DETAILED DESCRIPTION:
Participants in this study will participate in four visits; one screening visit and three study days.

Participants will be instructed to avoid strenuous exercise and alcohol intake two days prior to each experimental visit. Participants will arrive at the Department of Clinical Physiology and Nuclear Medicine after an overnight (>10 hours) fast (including coffee and medicine).

On all three study days, two peripheral venous catheters will be placed in the antecubital vein of each arm (one for the collection of blood samples and one for infusions). After two initial blood samples the infusion of either saline, glucagon or glucose will be started. The infusion rate of glucagon will be 10 ng/kg/min. The infusion rate of glucose will be adjustable, and adjusted to match the blood glucose levels achieved on the glucagon study day.

During the infusion of saline, glucagon or glucose a 18F-FDG PET/CT scan will be performed. The 18F-FDG PET/CT scan will be performed either in the beginning of the infusions (approximately 15-55 min after the start of infusion) (for participants in part C) or in the end of the infusions (approximately 150-190 min after the start of infusion) (for participants in part D).

ELIGIBILITY:
Inclusion Criteria:

* Age 55 to 70 years
* BMI under or equal to 30 kg/m2
* Capable of understanding the participant information and signing the consent form

Exclusion Criteria:

* Enrolment in other research projects that might interfere with the study
* Diabetes diagnosis (type 1 and 2)
* Use of medications which, in the opinion of the investigator, may jeopardise participant's safety or compliance with the protocol
* Diagnosis of psychiatric disorders, dementias, or any other neurological disorders that in the opinion of the investigator precludes compliance with the study protocol, evaluation of the results or represents an unacceptable risk for the participants safety
* Severe claustrophobia
* Impaired liver og kidney function
* Cardiac problems including any of the following:

  1. Classified as being in New York Heart Association (NYHA) class III or IV
  2. Angina pectoris (chest pain) within the last 6 months
  3. Acute myocardial infarction (heart attack) within last 2 years
* Inadequately treated blood pressure at screening defined as repeated resting blood pressure outside the range 90-150 mmHg for systolic and 50-100 mmHg for diastolic.
* Active or recent malignant disease
* Current or history of severe alcohol use or drug/chemical abuse as per investigator's judgement
* Any chronic disorders or severe diseases which, in the opinion of the investigator, might jeopardise participant's safety or compliance with the protocol

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Cerebral metabolic rate of glucose (CMRglc), acute effect (part C) | 15-55 minutes
  CMRglc is calculated based on the 18F-FDG PET/CT scan.

SECONDARY OUTCOMES:
Cerebral metabolic rate of glucose (CMRglc), later effect (part D) | 150-190 minutes
  CMRglc is calculated based on the 18F-FDG PET/CT scan.
Blood-brain glucose transfer capacity (Tmax), acute effect (part C) | 15-55 minutes
  Tmax is calculated based on the 18F-FDG PET/CT scan.
Blood-brain glucose transfer capacity (Tmax), later effect (part D) | 150-190 minutes
  Tmax is calculated based on the 18F-FDG PET/CT scan.
FDG net clearance (Ki), acute effect (part C) | 15-55 minutes
  Ki is calculated based on the 18F-FDG PET/CT scan.
FDG net clearance (Ki), later effect (part D) | 150-190 minutes
  Ki is calculated based on the 18F-FDG PET/CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai J Wewer Albrecthsen, MD PhD, Principal Investigator — Department of Clinical Biochemistry, Copenhagen University Hospital - Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark; Lisbeth J Marner, MD PhD, Study Chair — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Department of Clinical Physiology and Nuclear Medicine, Copenhagen University Hospital - Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark, Copenhagen, Denmark